CLINICAL TRIAL: NCT03619200
Title: FallSensing, a Multifactorial Screening Tool for Fall-risk in Community-dwelling Adults Aged 50 Years or Over
Status: Completed | Type: Observational
Sponsor: Anabela Correia Martins (Other)
Collaborators: Sensing Future Technologies (Other); Fraunhofer Portugal Research Center for Assistive Information and Communication Solutions (Other)
Responsible Party: Sponsor-Investigator, Anabela Correia Martins, Principal Investigator, Escola Superior de Tecnologia da Saúde de Coimbra
Organization: Escola Superior de Tecnologia da Saúde de Coimbra (Other)
Other Study IDs: 6/2017; POCI-01-0247-FEDER-003464 (Other Grant/Funding Number: co-funded by Portugal 2020, framed under the COMPETE 2020 and European Regional Development Fund (ERDF) from EU)
Record Dates: First submitted 2018-05-19; First posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Accidental Falls
Keywords: Primary prevention; Adults; Pressure platform; Inertial Sensors; Clinical Protocol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fallers: Participants who reported at least one fall in the 12-months follow-up period were categorized as "fallers".
- Non-Fallers: Participants who did not report any fall in the 12-months follow-up period were categorized as "non-fallers".

SUMMARY:
FallSensing screening tool is a technological solution for fall risk screening, including a software, a pressure platform and two inertial sensors. The screening includes questions about demographic and anthropometric data, health and lifestyle behaviors, a detailed explanation about procedures to accomplish six functional tests (Grip Strength, Timed Up and Go, 30 seconds Sit-to-Stand, Step test, 4 Stage Balance test "modified" and 10 meters Walking Speed) and three questionnaires concerning environmental home hazards, activities and participation profile related to mobility and self-efficacy for exercise.

DETAILED DESCRIPTION:
Variable: History of Fall (HoF) A fall can be defined as "an unexpected event in which the participant comes to rest on the ground, floor, or lower level" and "excludes coming to rest against furniture, wall, or other structure" .

The HoF within the previous 12 months will be determined by self-report, answering the question "Did you fall in the past 12 months? Yes-No". If the participant has fallen, it will be asked if the fall was outdoor or indoor, the reason of the fall (slip, stumble, loss of consciousness, dizziness, lower extremities weakness, no special reason and other), need of health services assistance, which health service (hospital, primary health care centre), hospitalization (how many days), activities limitation and restrictions on participation (how many days) and fractures occurrence (wrist or hand, hip, skull or spine, others).

Variable: History of falls after 12 months Participants will be prospectively followed for a 12-month period, via monthly phone calls, in order to record the falls occurrence. The rate of falls will be recorded from the day of inclusion until voluntary dropout, loss of phone contact or the end of the follow-up period (365 days later).

Variable: Fear of Falling (FoF) FoF is defined as "a lasting concern about falling that leads to an individual avoiding activities that he/she remains capable of performing".

Considering the negative influence of FoF, its existence will be assessed by self-report through the question "Are you afraid of falling? Yes - No".

Variable: Health Conditions There are certain conditions that can have a significant effect on fall rates among older adults, such as bladder incontinence, osteoarthritis, Parkinson's disease, cardiovascular accidents and conditions associated with cardiovascular disease, like hypertension.

The question "Do you have trouble seeing well or it has been past more than 2 years since your eyes have been tested?", once changes in visual acuity, development of cataracts, macular degeneration, glaucoma, and other conditions related to the aging process contribute to risk of falling.

Variable: Medication Older adults taking more than three or four medicines were found to be at increased risk of recurrent falls.

The number of medicines taken by each person was assessed by self-report through the question "Do you take 4 or more different medicines per day? Yes-No". The name of the medicines was also registered and they were identified according to their pharmaceutical group (benzodiazepines, antidepressants, antipsychotics, anti-inflammatory drugs, antihypertensive drugs and others drugs).

Variable: Sedentary Behavior In order to understand the community-dwelling adults' sedentary behavior by using a self-reported question, it was adopted the estimate measure of sedentariness calculated by Heseltine et al. (2015): "Do you spend over 4 hours seated, 5 days or more per week?".

Variable: Upper Extremities Assistance to Stand from a Chair The upper extremities assistance to stand from a chair was assessed through the question "Do you need assistance from the upper extremities to stand up from a chair? Yes-No", once it is assumed that is a sign of weak lower extremities muscles, a major reason for falling.

Variable: Living settings Since FoF is more frequent among older adults living alone, this protocol intends to assess the living settings through the question "Do you live alone? Yes-No".

Variable: Alcohol habits Regular alcohol consumption among older adults has been linked to impaired balance and postural hypotension, which has been associated with frequent falls.

The participants will be asked about their daily alcohol habits, "Do you drink alcohol every day? Yes-No".

Variable: Self-Perceived Health The self-perceived health (SPH) is considered a valid and reliable indicator of overall health status, a predictor of mortality and health services use.

SPH will be assessed by self-report through the question "In general, do you perceived your health as excellent, very good, good, sufficient or poor?"

Variable: Unintentional or involuntary weight loss The involuntary weight loss is one of the features that, simultaneously with others, can help to define a frailty phenotype.

The literature reveals an association between the frailty phenotype and the number of previous falls in older people. The participants will be asked if they had experienced a weight loss higher than ≥4,5kg or ≥5% of body weight during the previous 12 months.

Variable: Grip Strength The hand grip strength is significantly correlated with lower limb muscular strength, being a powerful predictor of disability, morbidity and mortality.

This test will be performed with the person seated on a standard chair without armrests, shoulder adducted and neutrally rotated, elbow flexed at 90 degrees, forearm neutral, wrist held between 0-15 degrees of ulnar deviation and with the arm not supported. A Jamar™ Hydraulic Hand Dynamometer will be settled at the second handle position, held with the dominant hand, and during the performance of the test will be presented vertically in line with the forearm. The test is performed only one time and the person is encouraged to exert her/his maximal grip strength for 5 seconds. The final score is measured in kilograms force (kgf). Normative data for this test are commonly analysed by gender, with males showing higher grip strength at all ages. A score below 15 kgf, for women, and 21 kgf, for men, identify those with higher risk of falling.

Variable:Timed Up and Go Timed Up and Go test (TUG) is used to assess dynamic balance during gait and transfers tasks, mobility and lower body strength. To perform this test, the person, wearing his/her regular footwear, is instructed to sit on a standard chair (chair height between 44 and 47 cm) with his/her back against the chair back, to stand up and walk straight for 3 meters as fast as possible, turn around, walk back and sit down. The person must stand up without help (cannot use the upper extremities for support), however if a walking aid is needed it should be placed next to the chair and can be used to perform the gait component of the test. The test is performed only one time, the timing begins at the instruction "go" and stops when the patient seats on the chair. A score higher than 10 seconds will indicate which community-dwelling older adults are more likely to be fallers.

Variable: 30 seconds Sit-to-Stand Lower body strength is a significant element to maintaining functional capacity in older adults, therefore its evaluation is critical. 30 seconds Sit-to-Stand (STS), being a simple and effective instrument for assessing lower body strength and identifying muscle weakness in community-dwelling older adults, is one of the most important functional evaluation clinical tests. The person is instructed to perform cycles of sits and stands up from a chair, as many times as possible over 30 seconds.

The person starts the test seated in the middle of the chair (chair height between 40 and 43,3cm), feet approximately shoulder-width apart and placed on the floor, and arms crossed by the wrists placed against the chest. The vocal instruction "go" sets the test´s beginning and if the participant completes more than halfway up at the end of 30 seconds it is counted as a full stand. Final score involves recording the number of stands a person can complete in 30 seconds. The normative levels for number of stands depends on age and gender.

Variable: Step Test The step test, was designed to assess the dynamic standing balance and reproduces lower-extremity motor control and coordination.

In order to perform the test, the person is asked to step on and off a block (7,5 cm height, 55 cm width, 35cm depth), placed against a wall, as many times as possible during 15 seconds. The whole foot is required to step onto the block and then return it fully to the ground. The total number of completed steps in 15 seconds is recorded. The patient is unsupported and should look straight forward, although investigator must stand close by for safety. In the case of patient overbalanced or need stabilization during the test, counting of steps stops and it is recorded the complete number of steps prior to overbalancing. This test is performed only for the dominant side, indicated by the person. A performance lower than 10 steps indicates higher risk of falling.

4 Stage Balance Test "Modified" Deficits in balance can lead to falls and fall related injuries, representing one of the most important intrinsic fall risk factors among older adults, being commonly assessed in this population.

The 4 Stage Balance Test "modified" is one of the tests available to evaluate balance. In order to complete this test, the person needs to progressively accomplish four different feet positions: side by side stance, semi-tandem stance (preferred foot forward with the instep of one foot touching the big toe of the other foot), tandem stance (one foot in front of the other, heel touching toe) and one legged stance (preferred leg for support).

The person is instructed to stand quietly on the pressure platform, arms along the body, neither with shoes or assistive devices. The positions must be held by 10 seconds each, without moving the feet, needing support, losing balance or touching the leg of support with the other leg, and must be performed with eyes open and then closed (excluding one legged stance position). The sequence will be side by side stance eyes open, side by side stance eyes closed, semi-tandem stance eyes open, semi-tandem stance eyes closed, tandem stance eyes open, tandem stance eyes closed and one leg stand eyes open. If the person failed to accomplish one of the test positions, the test finishes. The final score will be the number of positions successfully completed. The inability to complete 10 seconds in the tandem stance position, with eyes open, has been associated with higher risk of falling and mobility dysfunction.

10 meters Walking Speed Walking speed is the result of a complex interaction of multiple body structures and functions, such as lower extremity strength, proactive and reactive postural control, motor control or musculoskeletal condition. Accessing the gait speed (GS) as a screening tool can be useful to identify those at risk or in need of intervention, since the gait speed results are related to various health outcomes, like functional decline or fear of falling, besides GS can be a predictor of falls.

The performance of this test requires a 20 meters straight path, with 5 meters for acceleration, 10 meters for steady-state walking and 5 meters for deceleration. Markers are placed at the 0, 5, 15 and 20 meters positions of the path and the time to walk along the 5 and 15 meters is registered. The person is instructed to walk at his/her faster walking speed, without running, along the 20 meters path; an assistive device can be used if needed and the person should wear his/her regular footwear.

The range of normal walking speed is between 1,2 and 1,4 m/s, since it varies by age, gender and anthropometrics A value lower than 0,4m/s indicates a probability of needing an assistive device at home; 0,4 to 0,8 m/s is correlated with limited mobility; 0,8 to 1,25 m/s ambulation in the community with some risks; ≤ 1m/s subjects should start a program to reduce the risk of falling; ≥ 1,42 m/s is the safe streets crossing speed.

Questionnaires Self-efficacy for exercise The self-efficacy reflects the confidence that a person has to perform a certain behavior.

The self-efficacy for exercise is a 5-items scale intended to analyse the confidence that a person has to perform exercise according to five different emotional states, like feeling worried/having problems, feeling depressed, feeling tired, feeling tense and being busy.

Ratings are done using a 5-points Likert scale from 1 "not at all true" to 4 "completely true"; in between, 2 "slightly true" and 3 "moderately true".

Activities and Participation Profile related to Mobility (PAPM) The PAPM is an 18-items scale intended to improve understanding of the difficulties an individual experiences in performing certain daily activities in their natural environment. These activities can be conditioned by mobility and are related to the interactions and social relations, education, employment, money management, social and community life, influencing the active participation of any person as a full member of the society.

Ratings are done using a 5-points Likert scale from 0 "no limitation/restriction" to 4 "complete limitation/restriction". In between, 1 "mild limitation/restriction", 2 "moderate limitation/restriction" and 3 "severe limitation/restriction". Since some activities may not apply, not all activities may be rated. As a result, an individual's participation profile will be produced.

Home Safety Checklist for Fall Prevention The Home Safety Checklist for Fall Prevention is a 38-items scale intended to identify home hazards in each room of a person's home, namely hall and hallways, stairs, living/dining room, kitchen, bathroom, bedroom and outdoors.

Ratings are done using a 3 points scale from 0 "no risk", 1 "risk" to 99 "do not apply". A risk score is produced both to each room and for the home in general.

Statistical Analysis Statistical analysis will be performed using International Business Machines Statistical Package for the Social Sciences (IBM SPSS) (v.24) software. The sample size was calculated for infinite population for a 95% confidence interval and 5% margin of error, in order to assess the number of participants needed to consider a representative sample of Portuguese population (minimum of participants 385).

To perform the data analysis, the participants will be categorized as "fallers" (with one or more falls) and "non-fallers", according to the occurrence of falls during the 12 months follow-up period.

The statistical approach will be different according to the level of measurement for the variables. The descriptive analysis will determine mean and standard deviation for the quantitative variables and frequencies for the qualitative ones. Differences in the data between "fallers" and "non-fallers" will be analysed by Student t test for independent samples or Chi-square test. Binary logistic regression analysis will be performed to determine a model that allows the prediction of falls from the functional tests and other variables. Receiver-Operating Characteristic curves (ROC curve) analysis will be used to identify the best cut-off score that distinguishes "fallers" from "non-fallers". Sensitivity (percentage of "fallers" who were correctly identified), specificity (percentage of "non-fallers" that were correctly identified) and area under the receiver characteristic curve (AUC) of the model will be calculated for prediction of falls. A significance of 0.05 will be considered for all comparisons, except for the quality of adjustment of the regression models, obtained with the Hosmer and Lemeshow test, whose significance is considered for p≥0.05.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 50 years or over,
* Community-dweller
* independent to be standing and walking, with or without walking aids
* interest to participate in the study.

Exclusion Criteria:

* severe sensorial impairments (deafness or blindness)
* cognitive impairments which precludes the ability to comprehend the questionnaires and functional tests included in the screening protocol

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals are voluntarily recruited from several settings from the community, in different regions of continental Portugal, such as parish councils, physical therapy clinics, senior's universities and other facilities.
Sampling Method: Non-Probability Sample
Enrollment: 506 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

PRIMARY OUTCOMES:
History of Fall | Monthly for a 12 months period
  Falls occurrence in the 12 months follow up period. "Did you fall in the past month?"

SECONDARY OUTCOMES:
History of fall (Previous 12 months) | Day 0
  Falls occurrence 12 months prior to the screening. "Did you fall in the past 12 months?"
Fear of Falling | Day 0
  "Are you afraid of falling?"
Grip Strength | Day 0
  Kilogram-force
Timed Up and Go | Day 0
  seconds
30 seconds Sit-to-Stand | Day 0
  number of stands
Step Test | Day 0
  number of steps
4 Stage Balance Test "Modified" | Day 0
  last position accomplished
10 meters Walking Speed | Day 0
  meters per second
Self-efficacy for exercise | Day 0
  Score 5 to 20 points
Activities and Participation Profile related to Mobility (PAPM) | Day 0
  Classification: 0 "no limitation/restriction", 1 "mild limitation/restriction", 2 "moderate limitation/restriction", 3 "severe limitation/restriction", 4 "complete limitation/restriction"
Home Safety Checklist for Fall Prevention | Day 0
  Risk score from 0% (better) to 100% (worse), produced both to each room and for the home in general
Self-reported question on Urinary incontinence | Day 0
  "Do you leak urine when you laugh, cough, sneeze or lift weights?"
Self-reported question on Osteoarthritis | Day 0
  Have you ever been diagnosed with osteoarthritis?
Self-reported question on Parkinson's disease | Day 0
  Have you ever been diagnosed with Parkinson's disease?
Self-reported question on Osteoporosis | Day 0
  Have you ever been diagnosed with osteoporosis?
Self-reported question on High cholesterol | Day 0
  Have you ever been diagnosed with high cholesterol?
Self-reported question on Stroke | Day 0
  Have you ever suffered from a stroke?
Self-reported question on Heart attack | Day 0
  Have you ever suffered from a heart attack?
Self-reported question on Hypertension | Day 0
  Have you ever been diagnosed with hypertension?
Self-reported question on Diabetes | Day 0
  Have you ever been diagnosed with Diabetes?
Self-reported question on Vision impairment | Day 0
  "Do you have trouble seeing well or it has been past more than 2 years since your eyes have been tested?"
Self-reported question on Hearing problems | Day 0
  Do you have trouble hearing well?
Self-reported question on Medication | Day 0
  "Do you take 4 or more different medicines per day?"
Self-reported question on Sedentary Behavior | Day 0
  "Do you spend over 4 hours seated, 5 days or more per week?"
Self-reported question on Upper Extremities Assistance to Stand from a Chair | Day 0
  "Do you need assistance from the upper extremities to stand up from a chair?
Self-reported question on Living settings | Day 0
  "Do you live alone?"
Self-reported question on Alcohol habits | Day 0
  "Do you drink alcohol every day?"
Self-reported question on Self-Perceived Health | Day 0
  "In general, do you perceived your health as excellent, very good, good, sufficient or poor?"
Self-reported question on Unintentional or involuntary weight loss | Day 0
  The participants will be asked if they had experienced a weight loss higher than ≥4,5kg or ≥5% of body weight during the previous 12 months.